CLINICAL TRIAL: NCT01000857
Title: A Steady-state, Two-period Crossover Study to Compare the Pharmacokinetic Profile of Paroxetine After Repeated Daily Dosing of the Controlled-release Paroxetine Tablet (25 mg) With That of the Standard Immediate-release Paroxetine Tablet (20 mg) in Healthy Japanese Male Subjects
Brief Title: Repeat Dose Study of Controlled-Release Paroxetine Tablets and Immediate-Release Paroxetine Tablets in Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 112812
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Depressive Disorder
Keywords: controlled-release tablet; repeat dose; immediate-release tablet; paroxetine; safety; crossover; pharmacokinetics; steady-state; Japanese healthy male volunteers; tolerance
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label treatment with 2-period crossover design (Experimental): Group 1: Paroxetine CR 25 mg/day for 14 days / Paroxetine IR 20 mg/day for 14 days.
  Group 2: Paroxetine IR 20 mg/day for 14 days / Paroxetine CR 25 mg/day for 14 days.,
  PK results will be compared between the Paroxetine CR treatment period and the Paroxetine IR treatment period.
  Interventions: Drug: Paroxetine CR and Paroxetine IR

INTERVENTIONS:
Drug: Paroxetine CR and Paroxetine IR — Randomized, 2-period crossover repeat dosing of Paroxetine CR at 25 mg/day for 14 days and Paroxetine IR at 20 mg/day for 14 days in Japanese healthy male volunteers

SUMMARY:
The primary purpose of this study is to compare the steady-state pharmacokinetic profile of paroxetine CR (controlled-release) at the dosage of 25mg/day using the proposed final market tablet of CR 25mg in Japan with that of standard paroxetine IR(immediate-release ) at the dosage of 20mg/day using the currently marketed tablet of IR 20mg in Japan.

DETAILED DESCRIPTION:
This study is an open, randomized, repeat dose, two-period crossover design in Japanese healthy male volunteers. This clinical trial is designed primarily to compare the steady-state pharmacokinetic profile of paroxetine CR at the dosage of 25mg /day (25mg once daily for 14 days) using the proposed final market tablet of CR 25mg in Japan with that of paroxetine IR at the dosage of 20mg/day (20mg once daily for 14 days) using the currently marketed IR 20mg tablet in Japan, by the crossover oral repeat dosing manner.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese adult males between 20 and 64 years of age inclusive
* BMI 18.50 or higher and < 25.00 kg/m2, and bodyweight 50 kg or higher
* Non-smokers
* AST, ALT, ALP, gamma-GTP and total-bilirubin are below the upper limit of normal range
* QTc(B) interval <450 msec
* Able to attend all visits and complete the study
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* Any clinically relevant abnormality on the screening physical examination, vital signs, 12-lead ECG and/or clinical laboratory tests
* Medical history that is not considered as eligible for inclusion in this study by the investigator
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of asymptomatic gallstones)
* History of psychiatric disorder or suicide attempts or behaviours
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
* History of sensitivity to any of the paroxetine formulations, or components thereof
* Positive for urine drug screening
* Participation in another clinical study or post-marketing study in which the subject is or will be exposed to an investigational or a non-investigational product or device
* Participation in a clinical study or post-marketing study with an investigational or a non-investigational product or device within 4 months of preceding the first dose of study medication
* History of drug or other allergy, or idiosyncrasy, excluding a pollen allergy without current symptoms
* History of drug abuse, or current conditions of drug abuse or alcoholism
* History of regular alcohol consumption exceeding, on average, 14 drinks/week (1 drink = 150 mL of wine or 350 mL of beer or 45 mL of 80 proof distilled spirits) within 6 months of screening
* Use of prescription or no-prescription drugs, including vitamins, crude drug, herbal and dietary supplements (including St John's Wort) within 14 days prior to the first dose of study medication
* Unwillingness or inability to follow the procedures outlined in the protocol
* Consumption of grapefruit or grapefruit-containing products from 7 days prior to the first dose of study medication
* Positive for syphilis, HIV antibody and antigen, Hepatitis B surface antigen, Hepatitis C antibody or HTLV-1 antibody
* Donation of blood in excess of 400mL within the previous 4 months or 200mL within the previous 1 month to the first dose of study medication

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-11-05 (Actual); Primary Completion 2010-02-25 (Actual); Study Completion 2010-02-25 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of plasma paroxetine after 14-days repeat dosing of paroxetine CR at 25mg/day or paroxetine IR at 20mg/day | up to 96 hours after dosing on Day 14 of each treatment period of paroxetine CR or paroxetine IR

SECONDARY OUTCOMES:
Safety and tolerability in healthy Japanese male volunteers during and after the repeat dosing period of paroxetine CR or paroxetine IR | During the 14-days repeat dosing period and up to 96 hours after the last dose of paroxetine CR or paroxetine IR

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 112812 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112812?search=study&search_terms=112812#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 112812 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112812 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112812 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112812 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register